CLINICAL TRIAL: NCT07340749
Title: Cross-sectional Observational Study on the Impact of Neuromuscular Diseases on Quality of Life: Focus on Peripheral Neuropathies (Hereditary vs Inflammatory)
Brief Title: Quality of Life in Hereditary and Inflammatory Peripheral Neuropathies
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 26Neuro01
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hereditary and Inflammatory Peripheral Neuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Hereditary peripheral neuropathies: "WHODAS 2.0: Assesses daily functioning and disability across six domains: understanding, mobility, self-care, interpersonal relationships, domestic activities, and social participation.
  WHOQOL-BREF: Measures overall quality of life in four domains: physical, psychological, social relationships, and environment.
  MPT Questionnaire (SOTU and ATD PA): Evaluates participants' attitudes, perceptions, and professional practices in a specific organizational or educational context."
  Interventions: Other: WHODAS 2.0 questionnaire
- Patients with inflammatory peripheral neuropathies: "WHODAS 2.0: Assesses daily functioning and disability across six domains: understanding, mobility, self-care, interpersonal relationships, domestic activities, and social participation.
  WHOQOL-BREF: Measures overall quality of life in four domains: physical, psychological, social relationships, and environment.
  MPT Questionnaire (SOTU and ATD PA): Evaluates participants' attitudes, perceptions, and professional practices in a specific organizational or educational context."
  Interventions: Other: WHODAS 2.0 questionnaire

INTERVENTIONS:
Other: WHODAS 2.0 questionnaire — WHODAS 2.0: Assesses daily functioning and disability across six domains: understanding, mobility, self-care, interpersonal relationships, domestic activities, and social participation.
  WHOQOL-BREF: Measures overall quality of life in four domains: physical, psychological, social relationships, and environment.
  MPT Questionnaire (SOTU and ATD PA): Evaluates participants' attitudes, perceptions, and professional practices in a specific organizational or educational context.
  Other Names: WHOQOL BREF questionnaire; MPT Questionnaire (SOTU e ATD PA)

SUMMARY:
Neuromuscular diseases affect the nerves and muscles and can cause weakness, pain, fatigue, and difficulties in daily life. These problems may reduce independence, social participation, and overall quality of life.This observational study aims to evaluate the impact of peripheral neuropathies on quality of life. It focuses on two types of peripheral neuropathies: hereditary neuropathies, caused by genetic factors, and inflammatory neuropathies, caused by immune-related nerve damage. Adult patients with these conditions will be assessed at a single time point, without any change to their usual medical care. Participants will complete questionnaires about daily functioning, well-being, and quality of life. Some questions will also explore the use of assistive devices and supportive tools in everyday life.The study hypothesizes that peripheral neuropathies significantly affect quality of life and that this impact differs between hereditary and inflammatory forms. The results aim to improve understanding of patients' needs and support better, more personalized care."

ELIGIBILITY:
Inclusion Criteria:

* Clinical and paraclinical diagnosis compatible with hereditary or inflammatory peripheral neuropathy, confirmed by the investigating physicians (genetic results for HPN if available; clinical/electrophysiological criteria for IPN).
* Written informed consent.
* Ability to complete the questionnaires (or with the assistance of a caregiver if necessary, specifying the mode of assistance).

Exclusion Criteria:

* Legal incapacity (under guardianship or conservatorship).
* Moderate to severe cognitive impairment (e.g., MMSE < 27) preventing valid comprehension and completion of the questionnaires.
* Active cancer undergoing chemotherapy or radiotherapy (treatment likely to significantly alter quality of life in a non-specific way).
* Other acute serious medical conditions that could interfere with assessment, at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include two groups of patients. Group A will consist of 30 patients with hereditary peripheral neuropathy (e.g., Charcot-Marie-Tooth disease and other HPNs). Group B will include 30 patients with inflammatory peripheral neuropathy (e.g., acute or chronic inflammatory demyelinating polyneuropathies, autoimmune neuropathies).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (WHOQOL-BREF score) | At the inclusion
  Quality of life (WHOQOL-BREF score) at baseline (M0) in patients with hereditary peripheral neuropathy (HPN) and inflammatory peripheral neuropathy (IPN)

SECONDARY OUTCOMES:
Comparison of perceived quality of life | At the inclusion
  Comparison of perceived quality of life between HPN and IPN groups using WHOQOL-BREF scores
Association between functioning and quality of life | At the inclusion
  correlation between WHODAS 2.0 scores and WHOQOL-BREF scores.
Factors associated with impaired functioning and quality of life | At the inclusion
  identification of clinical or demographic variables linked to lower WHODAS 2.0 or WHOQOL-BREF scores.
Role of assistive technologies (MPT) | At the inclusion
  Evaluation of the impact or use of assistive technologies on functioning and quality of life.
Profile of limitations | At the inclusion
  Assessment using WHODAS 2.0 scores to describe functional limitations
Activity restrictions | At the inclusion
  Assessment using WHODAS 2.0 scores
Environmental factors | At the inclusion
  Assessment using WHODAS 2.0 scores

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France